CLINICAL TRIAL: NCT02016963
Title: An Open-Label Study to Evaluate the Immunogenicity and Safety of Raxibacumab (Human Monoclonal Antibody to B. Anthracis Protective Antigen) Administered in Healthy Subjects
Brief Title: An Open-label, Nonrandomized Study to Evaluate the Safety and Immunogenicity of Raxibacumab With Reinjection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry); Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGS1021-C1069; NCT03625479 (obsolete NCT alias)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Therapeutic Treatment of Inhalation Anthrax
Keywords: Monoclonal Antibody; Safety; Raxibacumab; HGS1021; Immunogenicity
MeSH Terms: interventions — raxibacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raxibacumab arm (Experimental): A maximum of 25 subjects (to include 3 evaluable female subjects) will receive a second dose of raxibacumab equal to that of the previous dose >= 4 months following the first dose.
  Interventions: Biological: Raxibacumab

INTERVENTIONS:
Biological: Raxibacumab — Raxibacumab will be supplied in 50 milliliter (mL) sterile, single-use vials containing 34.9 mL of liquid formulation per vial. Each vial contains 50 milligram (mg)/mL raxibacumab in 0.13 mg/mL citric acid, 2.8 mg/mL sodium citrate, 10 mg/mL sucrose, 18 mg/mL glycine, 0.2 mg/mL polysorbate 80, pH 6.5

SUMMARY:
This is an open-label study to evaluate the immunogenicity and safety of raxibacumab in healthy adult male and female subjects. Subjects who have received raxibacumab >= 4 months ago will be enrolled and dosed as follows: A maximum of 25 subjects (to include 3 evaluable female subjects) will receive a second dose of raxibacumab equal to that of the previous dose >= 4 months following the first dose. Subjects will remain in house from Day 0 until Day 1 and will be followed for 70 days after receiving the second dose of raxibacumab. Raxibacumab has been shown to provide improved survival in rabbit and monkey anthrax spore challenge studies. Preliminary data from our rabbit pivotal efficacy study showed significant survival benefit for raxibacumab over placebo. Exposure to anthrax and resulting clinical disease can occur more than once, especially in individuals who do not develop protective immunity. Hence, if clinically indicated for the treatment of anthrax, there may be a requirement for the repeat administration of raxibacumab. The rationale of the study is to evaluate the immunogenicity and safety of repeat administration of raxibacumab with a >= 4 month interval between dosing.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and treated with raxibacumab in another HGS protocol, >= 4 months ago.
* Male or female >= 18 and <= 64 years of age.
* Laboratory values that are Grade 0 by the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables. Subjects with laboratory values that are Grade 1 and are not considered clinically significant by the Principal Investigator may be enrolled following consultation with the Medical Monitor.
* A female subject is eligible to enter the study if she is: Not pregnant or nursing, Post menopausal, has had a hysterectomy, or documentation of sterility, Of child bearing potential (ie, woman with an intact uterus and ovaries and no documentation of oviductal or uterine dysfunction that would cause sterility).
* These women must have a negative blood pregnancy test at screening and on Day -1 prior to dosing and agree to 1 of the following: a)Complete abstinence from intercourse from the date of screening through the duration of follow-up, b)Consistent and correct use of 1 of the following medically accepted methods of birth control, in addition to a male partner who correctly uses a condom or is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subject from the date of screening through the duration of follow-up, implants of levonorgestrel; injectable progesterone; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progesterone only); double barrier method: condom, cervical cap or diaphragm with spermicidal agent; transdermal contraceptive patch.
* All males who are not sterile must agree to either abstain from intercourse or consistently and correctly use a condom while their female partner agrees to use 1 of the appropriate medically accepted methods of birth control listed above from the date of screening through the duration of follow-up.
* Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), comply with the study protocol procedures, and agree to return for the required study visits.

Exclusion Criteria:

* History or clinical evidence of significant, acute, or chronic diseases (ie, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological, or infectious diseases), which could confound the results of the study or put the subject at undue risk.
* Prior immunization with anthrax vaccine adsorbed (AVA), prior treatment with investigational anthrax therapies (other than raxibacumab >= 4 months ago), prior treatment for anthrax exposure, or a confirmed anthrax infection.
* History of Type I hypersensitivity reaction to food or drugs, intravenous (IV) contrast dye, or history of urticaria.
* Previous hypersensitivity to raxibacumab.
* Previous serious or Grade 3 or greater raxibacumab related adverse event (AE).
* Drug or alcohol addiction within the last 12 months. Subjects who have documented addiction free period of at least 12 months and in the clinical judgement of the investigator are not at risk for relapse may be enrolled in the study.
* Evidence of active or suspected malignancy or history of malignancy within the last 5 years (with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix).
* Participation in any other clinical trials of an investigational compound within 60 days of initiating study agent or refusal to refrain from participation during this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01-31 (Actual); Primary Completion 2008-05-31 (Actual); Study Completion 2008-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — Human Genome Sciences Inc.

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HGS1021-C1069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had received raxibacumab >= 4 months in another HGS study (study # HGS1021-C1064) prior to this study were eligible for enrollment in this study.
Groups:
- Raxibacumab: Participants received their second dose of raxibacumab 40 milligrams/kilogram (mg/kg) by intravenous (IV) infusion. Participants were treated with oral diphenhydramine 50 mg up to 60 minutes prior to infusion of raxibacumab.
Period: Overall Study
Arm/Group | Raxibacumab
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 13
  Black or African American | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed a Positive Anti-raxibacumab Antibody Response
Description: Number of participants who developed an positive anti-raxibacumab antibody response during the study were assessed.The antibody response to raxibacumab was assessed using a screening assay (i.e. by electrochemiluminescence counts). Positive samples would be further tested in an inhibition of binding assay to confirm the specificity of binding.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population : all participants who received 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. This includes worsening (eg, increase in frequency or severity) of pre-existing conditions. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Any AE | 8
  Any SAE | 0

3. Secondary Outcome: Number of Participants With Hematological Toxicities of the Indicated Grade
Description: Clinical hematological parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Leukocytosis, Grade 1 | 0
  Leukocytosis, Grade 2 | 0
  Leukocytosis, Grade 3 | 0
  Leukocytosis, Grade 4 | 0
  Leukopenia, Grade 1 | 5
  Leukopenia, Grade 2 | 0
  Leukopenia, Grade 3 | 0
  Leukopenia, Grade 4 | 0
  Lymphopenia, Grade 1 | 0
  Lymphopenia, Grade 2 | 1
  Lymphopenia, Grade 3 | 0
  Lymphopenia, Grade 4 | 0
  Neutropenia, Grade 1 | 2
  Neutropenia, Grade 2 | 0
  Neutropenia, Grade 3 | 0
  Neutropenia, Grade 4 | 0
  Hemoglobin, Grade 1 | 1
  Hemoglobin, Grade 2 | 0
  Hemoglobin, Grade 3 | 0
  Hemoglobin, Grade 4 | 0
  Platelet, Grade 1 | 0
  Platelet, Grade 2 | 0
  Platelet, Grade 3 | 0
  Platelet, Grade 4 | 0
  Prothrombin Time, Grade 1 | 0
  Prothrombin Time, Grade 2 | 0
  Prothrombin Time, Grade 3 | 0
  Prothrombin Time, Grade 4 | 1
  Partial Thromboplastin Time, Grade 1 | 0
  Partial Thromboplastin Time, Grade 2 | 1
  Partial Thromboplastin Time, Grade 3 | 0
  Partial Thromboplastin Time, Grade 4 | 0

4. Secondary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Hematological Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in hematological toxicities is presented. Clinical hematological parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Leukocytosis, any>=2-grade worsening | 0
  Leukopenia, any >=2-grade worsening | 0
  Lymphopenia, any>=2-grade worsening | 1
  Neutropenia, any >=2-grade worsening | 0
  Hemoglobin, any>=2-grade worsening | 0
  Platelet, any>=2-grade worsening | 0
  Prothrombin Time, any >=2-grade worsening | 1
  Partial Thromboplastin Time, any>=2grade worsening | 1

5. Secondary Outcome: Number of Participants With Liver Toxicities of the Indicated Grade
Description: Liver function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Aspartate amino transferase (AST), Grade 1 | 2
  AST, Grade 2 | 0
  AST, Grade 3 | 0
  AST, Grade 4 | 0
  Alanine amino transferase(ALT), Grade 1 | 1
  ALT, Grade 2 | 1
  ALT, Grade 3 | 0
  ALT, Grade 4 | 0
  Gamma-glutayl-transferase (GGT), Grade 1 | 0
  GGT, Grade 2 | 0
  GGT, Grade 3 | 0
  GGT, Grade 4 | 0
  Alkaline Phosphatase, Grade 1 | 0
  Alkaline Phosphatase, Grade 2 | 0
  Alkaline Phosphatase, Grade 3 | 0
  Alkaline Phosphatase, Grade 4 | 0
  Hyperbilirubinemia, Grade 1 | 0
  Hyperbilirubinemia, Grade 2 | 0
  Hyperbilirubinemia, Grade 3 | 0
  Hyperbilirubinemia, Grade 4 | 0

6. Secondary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Liver Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in liver toxicities is presented. Liver function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  AST, any>=2-grade worsening | 0
  ALT, any>=2-grade worsening | 1
  GGT, any>=2-grade worsening | 0
  Alkaline phosphatase, any>=2-grade worsening | 0
  Hyperbilirubinemia, any>=2-grade worsening | 0

7. Secondary Outcome: Number of Participants With Electrolyte Toxicities of the Indicated Grade
Description: Electrolyte function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Hypernatremia, Grade 1 | 0
  Hypernatremia, Grade 2 | 0
  Hypernatremia, Grade 3 | 0
  Hypernatremia, Grade 4 | 0
  Hyponatremia, Grade 1 | 2
  Hyponatremia, Grade 2 | 0
  Hyponatremia, Grade 3 | 0
  Hyponatremia, Grade 4 | 0
  Hyperkalemia, Grade 1 | 1
  Hyperkalemia, Grade 2 | 0
  Hyperkalemia, Grade 3 | 0
  Hyperkalemia, Grade 4 | 0
  Hypokalemia, Grade 1 | 0
  Hypokalemia, Grade 2 | 0
  Hypokalemia, Grade 3 | 0
  Hypokalemia, Grade 4 | 0
  Hypomagnesemia, Grade 1 | 0
  Hypomagnesemia, Grade 2 | 0
  Hypomagnesemia, Grade 3 | 0
  Hypomagnesemia, Grade 4 | 0
  Hypercalcemia, Grade 1 | 0
  Hypercalcemia, Grade 2 | 0
  Hypercalcemia, Grade 3 | 0
  Hypercalcemia, Grade 4 | 0
  Hypocalcemia, Grade 1 | 0
  Hypocalcemia, Grade 2 | 0
  Hypocalcemia, Grade 3 | 0
  Hypocalcemia, Grade 4 | 0
  Hypophosphatemia, Grade 1 | 1
  Hypophosphatemia, Grade 2 | 0
  Hypophosphatemia, Grade 3 | 0
  Hypophosphatemia, Grade 4 | 0

8. Secondary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Electrolyte Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in electrolyte toxicities is presented. Electrolyte function parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0.Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable. Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Hypernatremia, any>=2-grade worsening | 0
  Hyponatremia, any>=2-grade worsening | 0
  Hyperkalemia, any>=2-grade worsening | 0
  Hypokalemia, any>=2-grade worsening | 0
  Hypomagnesemia, any>=2-grade worsening | 0
  Hypercalcemia, any>=2-grade worsening | 0
  Hypocalcemia, any>=2-grade worsening | 0
  Hypophosphatemia, any>=2-grade worsening | 0

9. Secondary Outcome: Number of Participants With Other Chemistry Toxicities of the Indicated Grade
Description: Other chemistry parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Creatinine, Grade 1 | 0
  Creatinine, Grade 2 | 0
  Creatinine, Grade 3 | 0
  Creatinine, Grade 4 | 0
  Hypoalbuminemia, Grade 1 | 0
  Hypoalbuminemia, Grade 2 | 0
  Hypoalbuminemia, Grade 3 | 0
  Hypoalbuminemia, Grade 4 | 0
  Hyperuricemia, Grade 1 | 1
  Hyperuricemia, Grade 2 | 0
  Hyperuricemia, Grade 3 | 0
  Hyperuricemia, Grade 4 | 0
  Hyperglycemia, Grade 1 | 4
  Hyperglycemia, Grade 2 | 1
  Hyperglycemia, Grade 3 | 0
  Hyperglycemia, Grade 4 | 0
  Hypoglycemia, Grade 1 | 2
  Hypoglycemia, Grade 2 | 0
  Hypoglycemia, Grade 3 | 0
  Hypoglycemia, Grade 4 | 0
  Amylase, Grade 1 | 3
  Amylase, Grade 2 | 1
  Amylase, Grade 3 | 0
  Amylase, Grade 4 | 0

10. Secondary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Other Chemistry Toxicities
Description: The number of participants with at least a 2-grade worsening from Baseline in other chemistry toxicities is presented. Other clinical chemistry parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants
  Creatinine, any>=2-grade worsening | 0
  Hypoalbuminemia, any>=2-grade worsening | 0
  Hyperuricemia, any>=2-grade worsening | 0
  Hyperglycemia, any>=2-grade worsening | 1
  Hypoglycemia, any>=2-grade worsening | 0
  Amylase, any>=2-grade worsening | 0

11. Secondary Outcome: Number of Participants With Urinalysis Toxicities of the Indicated Grade
Description: Urinaysis parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants | 0

12. Secondary Outcome: Number of Participants With at Least a 2-grade Worsening From Baseline in Urinalysis Toxicities
Description: Urinalysis parameters were assessed using the modified Division of Microbiology and Infectious Diseases (DMID) toxicity tables, version 2.0. Grade 1 (Mild): Transient or mild discomfort (< 48 hours); no medical intervention or therapy required. Grade 2 (Moderate): Mild to moderate limitation in activity, some assistance may be needed; no or minimal medical intervention or therapy required. Grade 3 (Severe): Marked limitation in activity, some assistance usually required; medical intervention or therapy required, hospitalizations possible. Grade 4 (Life-threatening): Extreme limitation in activity, significant assistance required; significant medical intervention or therapy required, hospitalization or hospice care probable.Baseline is defined as the value of the variable measured at Day 0 prior to dosing.
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 70
Population: As-treated population
Measure: Number; unit: Participants
Arm/Group | Raxibacumab
Number analyzed (Participants) | 20
Participants | 0

13. Secondary Outcome: Mean Raxibacumab Concentration-time Following an IV Infusion Raxibacumab Dose
Description: Blood was collected from each participant at the selected times: pre-dose (Day 0), 0.00347 hours (Day 0), 0.3333 hours (Day 0), Day 1, Day 3, Day 7, Day 14, Day 21, Day 28, Day 42, and Day 56 post-dose. Serum specimens were analyzed for raxibacumab using a validated electrochemiluminescense-based assay. The individual serum raxibacumab concentration data were summarized by nominal collection time and treatment group using descriptive statistics
Time Frame: From the date of the dose administration of study agent for this study (Day 0) until Day 56
Population: As-treated population
Measure: Mean (Standard Deviation); unit: Micrograms/milliliter (µg/mL)
Groups:
- Raxibacumab IV: Participants received their second dose of raxibacumab 40 milligrams/kilogram (mg/kg) by intravenous (IV) infusion. Participants were treated with oral diphenhydramine 50 mg up to 60 minutes prior to infusion of raxibacumab.
Arm/Group | Raxibacumab IV
Number analyzed (Participants) | 20
Micrograms/milliliter (µg/mL)
  Pre-dose | 1.358 (1.879)
  0.00347 hr | 979.078 (147.543)
  0.3333 hr | 865.874 (122.602)
  Day 1 | 784.122 (118.680)
  Day 3 | 580.068 (94.776)
  Day 7 | 418.253 (62.350)
  Day 14 | 300.589 (41.689)
  Day 21 | 238.190 (39.515)
  Day 28 | 208.646 (44.802)
  Day 42 | 131.473 (44.308)
  Day 56 | 96.932 (46.637)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the time the first dose of study agent (Day 0) until Day 70.
Description: SAEs and non-serious AEs were collected in the as-treated population, comprised of all participants randomized to treatment who received one dose of study agent.
Arm/Group | Raxibacumab
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Raxibacumab (N=20)
Upper respiratory tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.